CLINICAL TRIAL: NCT05396885
Title: A Phase II Study of CART-ddBCMA for the Treatment of Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of Anitocabtagene-autoleucel in Relapsed or Refractory Multiple Myeloma (iMMagine-1)
Acronym: iMMagine-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Collaborators: Arcellx, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARC-112A
Record Dates: First submitted 2022-05-12; First posted 2022-05-31 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- anitocabtagene-autoleucel (Experimental): Single dose of 115±10 x 10e-6 CAR+ anitocabtagene-autoleucel cells infused intravenously
  Interventions: Biological: anitocabtagene-autoleucel

INTERVENTIONS:
Biological: anitocabtagene-autoleucel — Anitocabtagene-autoleucel-directed CAR T-cell therapy using a novel, synthetic binding domain, called a D-domain
  Other Names: CART-ddBCMA

SUMMARY:
A Phase II study of anitocabtagene-autoleucel (formerly CART-ddBCMA) for patients with relapsed or refractory multiple myeloma. Anitocabtagene-autoleucel is a BCMA-directed CAR-T cell therapy.

DETAILED DESCRIPTION:
This is a Phase II open-label study of anitocabtagene-autoleucel * in patients with relapsed or refractory multiple myeloma (MM). The study will have the following sequential phases: screening, enrollment, pre-treatment with lymphodepleting chemotherapy, treatment with anitocabtagene-autoleucel , and follow-up. If necessary, bridging therapy is allowed to control growth of MM disease while anitocabtagene-autoleucel is being manufactured.

Following a single infusion of anitocabtagene-autoleucel both safety and efficacy data will be assessed. Efficacy will be assessed monthly for the first 6 months, then quarterly up to 2 years, or upon patient relapse. The primary analysis will be conducted approximately 13 months after the final patient is dosed. This will allow approximately 12 months follow up from the time of the last observed response on study.

Long-term safety data will be collected under a separate long-term follow up study for up to 15 years per health authority guidelines.

*Anitocabtagene-autoleucel drug product consists of autologous T cells that have been genetically modified ex vivo to express a D-domain Chimeric Antigen Receptor (CAR), followed by a cluster of differentiation 8 (CD8) hinge and transmembrane region that is fused to the intracellular signaling domains for 4-1BB and CD3ξ, that specifically recognizes B-cell maturation antigen (BCMA). The active substance of anitocabtagene-autoleucel is CAR+ CD3+ T cells that have undergone ex vivo T-cell activation, gene transfer by replication-deficient lentiviral vector, and expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older and has capacity to give informed consent
2. Relapsed or refractory multiple myeloma treated with at least 3 prior regimens of systemic therapy including proteasome inhibitor, immunomodulatory drugs (IMiD) and anti-CD38 antibody and are refractory to the last line of therapy. For each line, 2 consecutive cycles are required unless the best response after 1 cycle was progressive disease.

   Note: IMWG criteria defines refractory disease as non-responsive to therapy or disease progression on or within 60 days of a therapy Note: Induction treatment with or without hematopoietic stem cell transplant and with or without maintenance is considered a single regimen
3. Documented measurable disease including at least one or more of the following criteria:

   1. Serum M-protein ≥1.0 g/dL
   2. Urine M-protein ≥200 mg/24 hours
   3. Involved serum free light chain ≥10 mg/dL with abnormal κ/λ ratio (i.e., >4:1 or <1:2)
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
5. Life expectancy >12 weeks
6. Adequate organ function defined as:

   1. Oxygen (O2) saturation ≥92% on room air
   2. Left Ventricular Ejection Fraction (LVEF) ≥45% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan
   3. Absolute neutrophil count (ANC) ≥1.0k/µl, platelet count (PLT)

      ≥50k/µl, [NOTE: Platelet transfusion not allowed within 14 days; filgrastim (or biosimilar) not allowed within 7 days, pegfilgrastim (or biosimilar) within 14 days]
   4. Creatinine clearance ≥45 mL/min min (as determined by the Cockgroft-Gault equation) and not on dialysis
   5. Aspartate transaminase (AST)/alanine transaminase (ALT) <3 x upper limits of normal (ULN)
   6. Total bilirubin <1.5 x ULN (allow 3x ULN for Gilbert's syndrome)
   7. Prothrombin time test (PTT), prothrombin time (PT)/international normalized ratio (INR) <1.5 x ULN, unless on a stable dose of anti-coagulant for a thromboembolic event (Subjects with any history of thromboembolic stroke; or history or Grade 2 (G2) or greater hemorrhage within one year are excluded)
7. Resolution of adverse events (AEs) from any prior systemic anticancer therapy, radiotherapy, or surgery to Grade 1 or baseline (except G2 alopecia and G2 sensory neuropathy)
8. Male and female participants of childbearing potential must agree to use highly effective methods of birth control through 12 months after the dose of study treatment
9. Willing to comply with and able to tolerate study procedures, including consent to participate in separate Long-term Safety Follow-up lasting up to 15 years per FDA guidance
10. Subject's leukapheresis product from non-mobilized cells is received and accepted for cell processing by manufacturing site. NOTE: Leukapheresis will be performed only after all other eligibility criteria are confirmed

Exclusion Criteria:

1. Plasma cell leukemia or history of plasma cell leukemia
2. Treatment with the following therapies as specified below

   1. Any prior systemic treatment for multiple myeloma within the 14 days prior to scheduled leukapheresis
   2. Receiving high-dose (e.g., >10 mg prednisone or equivalent) systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to leukapheresis
   3. Prior treatment with any gene therapy, gene-modified cellular immune-therapy, or T cell engager
   4. Prior B-cell maturation antigen (BCMA) directed therapy
   5. Autologous stem cell transplantation within 3 months prior to leukapheresis, or any prior allogeneic stem cell transplantation
3. Subjects with solitary plasmacytomas without evidence of other measurable disease are excluded
4. History of allergy or hypersensitivity to study drug components. Subjects with a history of severe hypersensitivity reaction to dimethyl sulphoxide (DMSO) are excluded
5. Contraindication to fludarabine or cyclophosphamide
6. Severe or uncontrolled intercurrent illness or laboratory abnormalities including

   1. Active bacterial, viral, or fungal infection requiring systemic treatment (isolated fever may not constitute active infection in and of itself, (e.g., related to disease)
   2. Symptomatic congestive heart failure (i.e., New York Heart Association stage III or IV)
   3. Unstable angina, arrhythmia, or myocardial infarction (MI) within 6 months prior to Screening
   4. Significant pulmonary dysfunction
   5. Uncontrolled thromboembolic events or recent severe hemorrhage (i.e., within one year)
   6. Any history of pulmonary embolism (PE) in the past 12 months or deep vein thrombosis (DVT) within three months of enrollment. Therapeutic dosing of anticoagulants (e.g., warfarin, low molecular weight heparin, Factor Xa inhibitors) is allowed for history of PE/DVT if greater than twelve and three months, respectively, from time of enrollment, and should be at a stable maintenance dose.
   7. Auto-immune disease requiring immunosuppressive therapy within the last 24 months
7. Seropositive for and with evidence of active hepatitis B or C infection at time of Screening, or HIV seropositive

   1. Subjects with a history of hepatitis B but have received antiviral therapy and have non-detectable viral DNA are eligible
   2. Subjects seropositive because of hepatitis B virus vaccine with no signs or active infection are eligible
   3. Subjects who had hepatitis C but have received antiviral therapy and show no detectable hepatitis C virus (HCV) viral RNA are eligible
8. Active central nervous system (CNS) involvement by malignancy
9. Any sign of active or prior CNS pathology including but not limited to history of epilepsy, seizure, paresis, aphasia, stroke, subarachnoid hemorrhage or CNS bleed, severe brain injury, dementia, cerebellar disease, Parkinson's disease, organic brain syndrome or psychosis
10. Active malignancy not related to myeloma that has required therapy in the last 3 years or is not in complete remission. Exceptions to this criterion include successfully treated non-metastatic basal cell or squamous cell skin carcinoma, or prostate cancer that does not require therapy.
11. Females who are pregnant or breastfeeding or females of childbearing potential not using an effective method of birth control
12. Subjects with any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in study (or full access to medical records) as written including follow up, the interpretation of data or place the subject at unacceptable risk
13. Any vaccine ≤ 6 weeks before leukapheresis and/or anticipation of the need for such a vaccine during the subject's participation in the study
14. Concurrent enrollment on another study using an investigational therapy for the treatment of RRMM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 24 Months
  ORR Per International Myeloma Working Group (IMWG) criteria, as assessed by an independent review committee (IRC)

SECONDARY OUTCOMES:
Stringent complete response (sCR) or complete response (CR) rate | 24 Months
  The proportion of participants in whom best response of sCR or CR,as assessed by an independent review committee (IRC) per by IMWG criteria
Overall Response Rate (ORR) of participants limited to three lines of prior treatment | 24 Months
  ORR per IMWG criteria, as assessed by an independent review committee (IRC), of participants limited to three lines of prior treatment
Duration of Response (DoR) | 24 Months
  DoR is defined as the time from the date of first documentation of response of PR or better per IMWG criteria after anitocabtagene-autoleucel infusion to the earlier of first documentation of disease progression per IMWG criteria or death
Very Good Partial Response (VGPR) Rate and Partial Response (PR) Rate | 24 Months
  The proportion of participants with best response of VGPR and PR, respectively, by IMWG criteria
Time to Initial Response | 24 months
  Time to initial response is defined as the measurement of time from the date of infusion of anitocabtagene-autoleucel to the date upon which the first IMWG response (i.e., PR or better) occurs
Progression Free Survival (PFS) | 24 Months
  PFS is defined as the measurement of time from the date of infusion of anitocabtagene-autoleucel to the date upon which the IMWG criteria for progressive disease or death occurs
Overall Survival (OS) | 24 Months
  OS is defined as the measurement of time (e.g., days or months) from the date of infusion of anitocabtagene-autoleucel to the date upon which death from any cause occurs
Safety Profile of anitocabtagene-autoleucel as assessed by incidence and severity of adverse events | 24 Months
  Summarization of adverse event (AE) terms, frequency, and severity using CTCAE version 5.0, the adverse events of special interest (AESIs), the serious adverse events (SAEs)
Pharmacokinetics of anitocabtagene-autoleucel | 24 Months
  Pharmacokinetics of anitocabtagene-autoleucel is defined as the using vector copy number (VCN) on peripheral mononuclear cells at defined timepoints. Quantification of anitocabtagene-autoleucel cells using vector copy number (VCN) on peripheral blood mononuclear cells
Anti-anitocabtagene-autoleucel Antibodies | 24 Months
  Proportion of participants who develop antibodies against anitocabtagene-autoleucel and the timing and titer of antibodies developed
Health Related Quality of Life (HRQoL) | 24 Months
  Measure the change in HRQoL pre- versus post-treatment with anitocabtagene-autoleucel
Minimal Residual Disease (MRD) negativity | 24 Months
  The proportion of participants that are MRD negative (i.e., no measurable tumor cells in at least 105 cells isolated from the bone marrow) from the efficacy evaluable (EE) population and from the MRD evaluable population (i.e., those participants with baseline sample allowing MRD calibration)
Time to Progression (TTP) | 24 Months
  TTP is defined as the measurement of time from date of anitocabtagene-autoleucel infusion to first documented IRC assessed progression using IMWG criteria or death due to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Arcellx, Inc., Study Director — Arcellx, Inc.
Locations (18):
- United States (18):
  - HonorHealth Cancer Transplant Institute, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Levine Cancer Institute, Charlotte, North Carolina
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT05396885